CLINICAL TRIAL: NCT06819384
Title: Effects of Movement Pattern Training Versus Proprioceptive Neuromuscular Training on Pain Range of Motion Flexibility and Kick Distance in Footballers With Groin Pain
Brief Title: Effects of Movement Pattern Training Versus Proprioceptive Neuromuscular Training in Footballers With Groin Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0403
Record Dates: First submitted 2024-11-18; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sports Physical Therapy
Keywords: Groin; Hip; Movements; Physiotherapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment randomized control design
Who Masked: Participant
Masking Description: Single (Participant) the participants are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Pattern Training (Experimental): The group A Comprises 18 participants and will perform Movement Pattern Training 2set each set 20 repition lasting for eight weeks.
  Interventions: Other: Movement Pattern Training
- propioceptive neuromuscular facilitation (Experimental): The group B Comprises 18 participants and will perform propioceptive neuromuscular facilitation 2set each set 20 repition lasting for eight weeks.
  Interventions: Other: propioceptive neuromuscular facilitation

INTERVENTIONS:
Other: Movement Pattern Training — The group A Movement Pattern Training 2set each set 20 repition lasting for eight weeks.
  Arms: Movement Pattern Training
Other: propioceptive neuromuscular facilitation — The group B propioceptive neuromuscular facilitation 2set each set 20 repition lasting for eight weeks.
  Arms: propioceptive neuromuscular facilitation

SUMMARY:
Effects Of Movement Pattern Training Versus Proprioceptive Neuromuscular Facilitation On Pain Range Of Motion Flexibility and Kick Distance Among Footballers With Groin Pain.

DETAILED DESCRIPTION:
According to the literature, due to the small number of PT studies on elite athletes (compared with the number of studies on general athletes), it is necessary to further understand whether PT can also benefit this group and accurately test the sports science equipment to facilitate the planning of accurate training courses.There is limited number of studies that have investigated comparative effects of pattern training and propiocetive neuro muscular facilitation..Also, there was no study found that Effects Of Movement Pattern Training Versus Proprioceptive Neuromuscular Facilitation On Pain Range Of Motion Flexibility and Kick Distance Among Footballers With Groin Pain.

ELIGIBILITY:
Inclusion Criteria:

* History of groin or adductor strain Patient Neurological involvement that influenced coordination or balance
* Male players,groin pain during or after the game
* groin pain > 8 weeks.
* Tenderness on palpation.
* pain during hip adduction with resistance
* Willingness to participate in the research

Exclusion Criteria:

* Subjects with urinary tract infection
* Lower limb fractures,
* metastasis
* Spinal pathology,
* hip joint osteoarthritis
* Inguinal pain(2).

Ages: 15 Years to 41 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
International Hip Outcome Tool | 8 weeks
  Overall iHOT-33 and iHOT-12 scores were calculated as the mean visual analog scale score for the individual items for each questionnaire for each patient)
Sit And Reach Flexibility Test. | 8 weeks
  The sit and reach test is a common measure of flexibility, and specifically measures the flexibility of the lower back and hamstring muscles.sit and reach box (or alternatively a ruler can be used, and a step or box)
Hip Rotation (Goniometer) | 8 weeks
  Hip Internal and External Rotation Range of motions will be measured
Kicking For Distance | 8 weeks
  Measuring Tapes will be used to measure the kick distance

CONTACTS AND LOCATIONS:
Overall Officials: Awais ul Mustafa, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Academy, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bialosky JE, Beneciuk JM, Bishop MD, Coronado RA, Penza CW, Simon CB, George SZ. Unraveling the Mechanisms of Manual Therapy: Modeling an Approach. J Orthop Sports Phys Ther. 2018 Jan;48(1):8-18. doi: 10.2519/jospt.2018.7476. Epub 2017 Oct 15. PMID 29034802
- [Background] Mastenbrook MJ, Commean PK, Hillen TJ, Salsich GB, Meyer GA, Mueller MJ, Clohisy JC, Harris-Hayes M. Hip Abductor Muscle Volume and Strength Differences Between Women With Chronic Hip Joint Pain and Asymptomatic Controls. J Orthop Sports Phys Ther. 2017 Dec;47(12):923-930. doi: 10.2519/jospt.2017.7380. Epub 2017 Oct 9. PMID 28992772
- [Background] Palaniappan R, Harris MD, Steger-May K, Bove AM, Fitzgerald GK, Clohisy JC, Harris-Hayes M. Comparison Between Movement Pattern Training and Strengthening on Kinematics and Kinetics in Patients With Chronic Hip-Related Groin Pain. J Appl Biomech. 2023 Nov 8;40(2):91-97. doi: 10.1123/jab.2022-0304. Print 2024 Apr 1. PMID 37939703
- [Background] McCrory P, Bell S. Nerve entrapment syndromes as a cause of pain in the hip, groin and buttock. Sports Med. 1999 Apr;27(4):261-74. doi: 10.2165/00007256-199927040-00005. PMID 10367335
- [Background] Rivadulla AR, Gore S, Preatoni E, Richter C. Athletic groin pain patients and healthy athletes demonstrate consistency in their movement strategy selection when performing multiple repetitions of a change of direction test. J Sci Med Sport. 2020 May;23(5):442-447. doi: 10.1016/j.jsams.2019.12.011. Epub 2019 Dec 17. PMID 31870678
- [Background] King MG, Schache AG, Semciw AI, Middleton KJ, Heerey JJ, Kemp JL, Sritharan P, Scholes MJ, Mentiplay BF, Crossley KM. Lower-limb work during high- and low-impact activities in hip-related pain: Associations with sex and symptom severity. Gait Posture. 2021 Jan;83:1-8. doi: 10.1016/j.gaitpost.2020.09.025. Epub 2020 Sep 29. PMID 33032182
- [Background] Kemp JL, Mosler AB, Hart H, Bizzini M, Chang S, Scholes MJ, Semciw AI, Crossley KM. Improving function in people with hip-related pain: a systematic review and meta-analysis of physiotherapist-led interventions for hip-related pain. Br J Sports Med. 2020 Dec;54(23):1382-1394. doi: 10.1136/bjsports-2019-101690. Epub 2020 May 6. PMID 32376673
- [Background] Palsson A, Kostogiannis I, Ageberg E. Physical impairments in longstanding hip and groin pain: Cross-sectional comparison of patients with hip-related pain or non-hip-related groin pain and healthy controls. Phys Ther Sport. 2021 Nov;52:224-233. doi: 10.1016/j.ptsp.2021.09.011. Epub 2021 Sep 30. PMID 34628337
- [Background] Melugin HP, Hale RF, Zhou J, LaPrade M, Bernard C, Leland D, Levy BA, Krych AJ. Risk Factors for Long-term Hip Osteoarthritis in Patients With Femoroacetabular Impingement Without Surgical Intervention. Am J Sports Med. 2020 Oct;48(12):2881-2886. doi: 10.1177/0363546520949179. Epub 2020 Aug 21. PMID 32822223
- [Background] Chang A, Ly NK, Varacallo MA. Piriformis Injection. 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448193/ PMID 28846327